CLINICAL TRIAL: NCT03553628
Title: Using a Mouthwash Containing Propolis, Clove Oil and Chlorhexidine to Improve the Caries Risk of High Risk Patients: Randomized Clinical Trial
Brief Title: Using a Mouthwash Containing Propolis, Clove Oil and Chlorhexidine to Improve the Caries Risk of High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moataz Gamal Ali Abdul-Maksoud Konsouh (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Moataz Gamal Ali Abdul-Maksoud Konsouh, Master Candidate at Conservative Department, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: oper252215
Record Dates: First submitted 2018-05-30; First posted 2018-06-12 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Caries, Dental; Risk Reduction
Keywords: dental caries; propolis; chlorhexidine; clove oil; bee wax
MeSH Terms: conditions — Dental Caries; Risk Reduction Behavior | interventions — Chlorhexidine; Propolis

STUDY DESIGN:
Intervention Model Description: A total of 64 patients will be assigned in this study. Patients will be randomly divided into two groups according to type of mouthwash (A) where group A1 patients will use chlorhexidine mouthwash as control group while group A2 patients will use chlorhexidine with propolis and clove oil mouthwash as intervention group with 32 patients in each group. Each group will be further divided into two groups according to times of application (T) where T1 represents patients using the mouthwash once daily for one week every month for 6 months and T2 where patients will use the mouthwash twice daily for one week every month for 6 months with 16 patients in each subgroup.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation of mouthwash and times of applications to groups will be done through sealed opaque sequentially numbered containers to ensure absolute concealment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chlorhexidine Once Daily (Active Comparator): Chlorhexidine HCL 0.12% mouthwash to be used once daily for one week each month for six months
  Interventions: Other: Chlorhexidine mouthwash
- Chlorhexidine Twice Daily (Active Comparator): Chlorhexidine HCL 0.12% mouthwash to be used twice daily for one week each month for six months
  Interventions: Other: Chlorhexidine mouthwash
- Propolis Once Daily (Experimental): Chlorhexidine Gluconate 0.12% with Propolis 1% and Clove Oil 1% mouthwash to be used once daily for one week each month for six months
  Interventions: Other: Chlorhexidine, Propolis and Clove Oil mouthwash
- Propolis Twice Daily (Experimental): Chlorhexidine Gluconate 0.12% with Propolis 1% and Clove Oil 1% mouthwash to be used twice daily for one week each month for six months
  Interventions: Other: Chlorhexidine, Propolis and Clove Oil mouthwash

INTERVENTIONS:
Other: Chlorhexidine, Propolis and Clove Oil mouthwash — Chlorhexidine Gluconate 0.12% with Propolis 1% and Clove Oil 1% mouthwash
  Arms: Propolis Once Daily; Propolis Twice Daily
Other: Chlorhexidine mouthwash — Chlorhexidine HCL 0.12% mouthwash
  Arms: Chlorhexidine Once Daily; Chlorhexidine Twice Daily

SUMMARY:
This study is conducted to determine if using a mouthwash containing propolis, clove oil and chlorhexidine will improve the caries risk of high risk patients in comparison to using a mouthwash containing chlorhexidine only.

DETAILED DESCRIPTION:
A total of 64 patients will be assigned in this study. Patients will be randomly divided into two groups according to type of mouthwash (A) where group A1 patients will use chlorhexidine mouthwash as control group while group A2 patients will use chlorhexidine with propolis and clove oil mouthwash as intervention group with 32 patients in each group. Each group will be further divided into two groups according to times of application (T) where T1 represents patients using the mouthwash once daily for one week every month for 6 months and T2 where patients will use the mouthwash twice daily for one week every month for 6 months with 16 patients in each subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be over 18 years of age.
* Patients should be with high caries risk assessment.

Exclusion Criteria:

* Patients with a compromised medical history.
* Severe or active periodontal disease.
* Patients with a diseased salivary gland
* History of allergies or other adverse reactions to chlorhexidine, propolis, bee stings, or clove
* Patients on any antibiotics during the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Caries Risk Assessment | 6 month
  Patient caries risk assessment will be measured using the cariogram model

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad A Ezzat, Ph.D., Study Director — Cairo University
Locations (1):
- Conservative Dentistry Department Out-Patient Clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alian AY, McNally ME, Fure S, Birkhed D. Assessment of caries risk in elderly patients using the Cariogram model. J Can Dent Assoc. 2006 Jun;72(5):459-63. PMID 16772072
- [Background] Autio-Gold J. The role of chlorhexidine in caries prevention. Oper Dent. 2008 Nov-Dec;33(6):710-6. doi: 10.2341/08-3. PMID 19051866
- [Background] Duailibe SA, Goncalves AG, Ahid FJ. Effect of a propolis extract on Streptococcus mutans counts in vivo. J Appl Oral Sci. 2007 Oct;15(5):420-3. doi: 10.1590/s1678-77572007000500009. PMID 19089172
- [Background] Eley BM. Antibacterial agents in the control of supragingival plaque--a review. Br Dent J. 1999 Mar 27;186(6):286-96. doi: 10.1038/sj.bdj.4800090. PMID 10230103
- [Background] Grossman, E., Retter, G., Sturzenberger, O. P., Rosa, M. D. La, Dickinson, T. D., Ferretti, G. A., … Meckel, A. H. (1986). Six-month Study of the Effects of a Chlorhexidine Mouthrinse on Gingivitis in Adults. Journal of Periodontal Research, 33-43.
- [Background] Hegde KS, Bhat SS, Rao A, Sain S. Effect of Propolis on Streptococcus mutans Counts: An in vivo Study. Int J Clin Pediatr Dent. 2013 Jan;6(1):22-5. doi: 10.5005/jp-journals-10005-1180. Epub 2013 Apr 26. PMID 25206182
- [Background] Kim MJ, Kim CS, Kim BH, Ro SB, Lim YK, Park SN, Cho E, Ko JH, Kwon SS, Ko YM, Kook JK. Antimicrobial effect of Korean propolis against the mutans streptococci isolated from Korean. J Microbiol. 2011 Feb;49(1):161-4. doi: 10.1007/s12275-011-1002-8. Epub 2011 Mar 3. PMID 21369995
- [Background] Liberio SA, Pereira AL, Araujo MJ, Dutra RP, Nascimento FR, Monteiro-Neto V, Ribeiro MN, Goncalves AG, Guerra RN. The potential use of propolis as a cariostatic agent and its actions on mutans group streptococci. J Ethnopharmacol. 2009 Aug 17;125(1):1-9. doi: 10.1016/j.jep.2009.04.047. Epub 2009 May 5. PMID 19422903
- [Background] Anauate Netto C, Marcucci MC, Paulino N, Anido-Anido A, Amore R, de Mendonca S, Borelli Neto L, Bretz WA. Effects of typified propolis on mutans streptococci and lactobacilli: a randomized clinical trial. Braz Dent Sci. 2013 Apr 1;16(2):31-36. doi: 10.14295/bds.2013.v16i2.879. PMID 24494174
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464